CLINICAL TRIAL: NCT04009330
Title: Clinical Evaluation of a POC Assay to Identify Phenotypes in the Acute Respiratory Distress Syndrome
Brief Title: Clinical Evaluation of a Point of Care (POC) Assay to Identify Phenotypes in the Acute Respiratory Distress Syndrome
Acronym: PHIND
Status: Active, not recruiting | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: Northern Ireland Clinical Trials Unit (Other); Innovate UK (Other Government)
Responsible Party: Principal Investigator, DannyMcAuley, Professor, Queen's University, Belfast
Other Study IDs: B19/06
Record Dates: First submitted 2019-05-15; First posted 2019-07-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: hyper and hypo-inflammatory; Phenotypes; POC (point of care)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples to be retained are: Li heparin plasma, Na3citrate plasma, Serum, Pax-Gene DNA, PBMC, Pax-Gene RNA and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Adults in the Intensive Care Setting: Adults in the Intensive Care Setting
  Interventions: Diagnostic Test: POC Assay

INTERVENTIONS:
Diagnostic Test: POC Assay — Interventions:
  Blood Baseline - up to 40ml Day 3 - up to 40ml
  Urine Baseline - 10ml Day 3 - 10ml
  Study population:
  Adults (18 plus) in ICU units diagnosed with ARDS.

SUMMARY:
Patients prospectively classified to the hyper-inflammatory ARDS phenotype on the basis of clinical characteristics and a novel POC biomarker assay will have worse clinical outcomes than the hypo-inflammatory phenotype.

Study Aim

The purpose of this project is to prospectively identify hyper- and hypo-inflammatory phenotypes in patients with ARDS and determine clinical outcomes associated with each phenotype.

The primary objective of this study is to assess the clinical outcomes in patients with ARDS according to their prospectively defined inflammatory phenotype determined using a POC assay.

Results of group allocation will be blinded to clinical and research staff until database lock.

Secondary Objectives

The secondary objectives of this study are to:

(i) Assess the agreement of the phenotype allocation using the POC assay and the clinical study dataset.

(ii) Assess the stability of phenotype allocation over time

(iii) To test feasibility of delivering a POC assay in the NHS intensive care setting.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is an inflammatory condition that results in severe respiratory failure and the need for mechanical ventilation. It is a syndrome with significant global burden and accounts for approximately 24% of mechanically ventilated patients in intensive care units. It is estimated to account for approximately 75000 deaths annually in the USA alone.

Despite decades of research, mortality due to ARDS remains high at 35-46%, with increasing mortality in patients with more severe lung injury. ARDS survivors have significant long term comorbidity with reduced quality of life even 5 years after disease resolution. Various pharmacological agents such as β2 agonists, statins, keratinocyte growth factor and aspirin have been investigated as potential therapies to prevent or treat ARDS, however to date there is no effective pharmacological therapy for ARDS and current treatment strategy is largely supportive.

One reason for the lack of specific pharmacological therapy is likely due to the clinical and biological heterogeneity. It is essential to rapidly identify patients with specific therapy responsive traits to improve our chance of identifying a specific therapy.

Rationale for the Study

ARDS phenotypes have different outcomes and response to therapy.

The clinical and biological heterogeneity in ARDS makes it essential to identify homogenous phenotypes when investigating potential therapies.

A retrospective analysis of the clinical and biological data-set collected as part of two large multicentre studies (ARMA and ALVEOLI) using latent class analysis has identified at least two ARDS phenotypes. Furthermore these two phenotypes could be differentiated using a parsimonious data-set including the presence of shock, metabolic acidosis and a higher inflammatory status (IL-6 and sTNFr1). The hyper-inflammatory phenotype demonstrated significantly worse outcomes when compared to the hypo-inflammatory phenotype with higher mortality and less ventilator free and organ failure free days. In the ALVEOLI study, where low PEEP was compared to high PEEP strategy, the two phenotypes demonstrated a differential response to PEEP suggesting the potential for using this phenotypic classification in identifying a therapy responsive trait.

In addition, in a secondary analysis of the HARP-2 study, a multicentre study investigating the potential of simvastatin as an anti-inflammatory therapy for ARDS, the presence of a hyper- and hypo-inflammatory phenotype was confirmed. The hyper-inflammatory phenotype had a higher 28 day mortality, fewer ventilator free days and organ failure free days. Survival of patients classified as hyper-inflammatory and randomised to simvastatin was improved.

Implementation of a precision medicine approach to identify patients with a therapy response trait is crucial to identify specific therapies to prevent or treat ARDS. Development of a Point of Care (POC) assay for IL-6 and sTNFr1 for prospective confirmation of the inflammatory phenotypes using the parsimonious data-set in patients with ARDS will support a precision medicine approach for this condition.

A POC assay will support precision medicine for ARDS

Studies that show no benefit from an intervention could occur as a result of a variety of reasons including a) the intervention was ineffective, b) the study design was poor or c) patient heterogeneity. Reduction of patient heterogeneity to identify patients with common biological processes will enable the selection of patients with a higher likelihood of therapy response in clinical studies. The identification and institution of therapy for critically ill patients with ARDS needs to occur rapidly in view of the nature of the disease and development of an accurate POC assay is likely to be an essential component in the discovery of effective therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is receiving mechanical ventilation or high flow nasal oxygen (HFNO)
2. ARDS as defined by the Berlin definition (Ranieri et al.) a) Onset within 1 week of identified insult b) Within the same 24-hour time period: i. Hypoxic respiratory failure (PaO2/ FiO2 ratio ≤ 40kPa on PEEP ≥ 5 cmH20*) ii. Bilateral infiltrates consistent with pulmonary oedema not explained by another pulmonary pathology iii. Respiratory failure not fully explained by cardiac failure or fluid overload

The time of onset of ARDS is when the last ARDS criterion is met.

*PEEP assumed ≥ 5 cmH20 if on HFNO.

Exclusion Criteria:

1. Age <18 years of age
2. More than 48 hrs after onset of ARDS
3. Receiving ECMO at the time of recruitment
4. Treatment withdrawal imminent within 24 hours
5. DNAR (Do Not Attempt Resuscitation) order (excluding advance directives) in place
6. Declined consent
7. Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS in the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is mortality at 60 days in the hyper-inflammatory and hypo-inflammatory phenotypes in patients with ARDS. | 60 days
  The primary outcome is mortality at 60 days in the hyper-inflammatory and hypo-inflammatory phenotypes in patients with ARDS.

SECONDARY OUTCOMES:
Difference in time to extubation | 60 days
  Difference in time to extubation
Intubation rate in patients on HFNO | 60 days
  Intubation rate in patients on HFNO
Reintubation Rate | 60 days
  Reintubation Rate
Number of ventilator free days at day 28 | 28 days
  Number of ventilator free days at day 28
Number of days on ventilation | 60 days
  Number of days on ventilation
Length of ICU stay | 60 days
  Length of ICU stay
Length of hospital stay | 60 days
  Length of hospital stay
Mortality at day 28 | 28 days
  Mortality at day 28
Agreement of phenotype classification using a POC assay and standard laboratory based assays. | Day 1 and day 3
  Agreement of phenotype classification using a POC assay and standard laboratory based assays.
Agreement of phenotype classification using a POC assay and the clinical study dataset. | 2 Years
  Agreement of phenotype classification using a POC assay and the clinical study dataset.
Agreement of phenotype classification between day 1 and day 3. | Day 1 and Day 3
  Agreement of phenotype classification between day 1 and day 3.
Frequency of assay technical failure rate will be used to determine the feasibility of delivering a POC assay in NHS intensive care setting. | 2 years
  Frequency of assay technical failure rate will be used to determine the feasibility of delivering a POC assay in NHS intensive care setting.

CONTACTS AND LOCATIONS:
Overall Officials: Professor D McAuley, Principal Investigator — Queens University Belfast
Locations (22):
- St Vincents Hospital, Dublin, Ireland, Ireland
- United Kingdom (21):
  - University Hospital Birmingham, Birmingham, England
  - Royal Blackburn Hospital, Blackburn, England
  - Royal Liverpool University Hospital, Liverpool, England
  - University College London, London, England
  - Guys and St Thomas Hospital, London, England
  - Kings College Hospital, London, England
  - Wythenshawe Hospital, Manchester, England
  - Manchester Royal Infirmary, Manchester, England
  - Freemans Hospital, Newcastle upon Tyne, England
  - Nottingham University Hospital, Nottingham, England
  - Royal Berkshire Hospital, Reading, England
  - Sunderland Royal, Sunderland, England
  - Royal Cornwall Hospital, Truro, England
  - Edinburgh Royal Infirmary, Edinburgh, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - University Hospital of Wales, Cardiff, Wales
  - Royal Gwent Hospital, Newport, Wales
  - Royal Victoria Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Imperial College London, London
  - Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Following the publication of the primary and secondary outcomes there may be scope to conduct additional analyses on the data collected. In such instances formal requests for data will need to be made in writing to the CI via the Northern Ireland Clinical Trials Unit, who will discuss this with the sponsor.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following the publication of the primary and secondary outcomes.
Access Criteria: Formal requests for data will need to be made in writing to the CI via the Northern Ireland Clinical Trials Unit, who will discuss this with the sponsor.
URL: http://www.nictu.hscni.net/PHIND

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452